CLINICAL TRIAL: NCT04816552
Title: Water, Sanitation, and Hygiene Mobile Health Messages as an Innovative Tool to Facilitate Behavior Change (CHoBI7 Program)
Brief Title: Water, Sanitation, and Hygiene Mobile Health Messages as an Innovative Tool to Facilitate Behavior Change
Acronym: CHoBI7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9255; IRB00009255 (Other: JHSPH IRB)
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHoBI7 mHealth program Arm (Experimental): The first arm will receive the CHoBI7 mHealth program and a general message on oral rehydration solution (ORS) (CHoBI7 mHealth program Arm) .
  Interventions: Behavioral: CHoBI7 mHealth program Arm; Behavioral: general message on oral rehydration solution (ORS)
- Standard Recommendation Arm (Active Comparator): The second arm will serve as a Control Arm and only receive a general message on oral rehydration solution (ORS).
  Interventions: Behavioral: general message on oral rehydration solution (ORS)

INTERVENTIONS:
Behavioral: CHoBI7 mHealth program Arm — We will start delivery of this intervention with a pictorial module delivered in the home during two 30 minute visits on cholera transmission and prevention after enrollment. Households will be provided a handwashing station, a covered water vessel, and chlorine tablets. Households will then receive the CHoBI7 WASH mHealth program voice and text messages on handwashing with soap and water treatment bi-weekly.
  Arms: CHoBI7 mHealth program Arm
Behavioral: general message on oral rehydration solution (ORS) — general message on oral rehydration solution (ORS)

SUMMARY:
Develop a scalable approach for delivering water, sanitation, and hygiene (WASH) messages to households in areas with confirmed cholera patients in Dhaka, Bangladesh. This will be done by conducting formative research through in-depth interviews, focus group discussions, and intervention planning workshops with households in areas with confirmed cholera patients and government officials to identify perceptions of WASH behaviors and to inform the development of a mobile health intervention (mHealth) for this population. This intervention approach will then be piloted in a subset of households, and revised according to feedback. Then the investigators will conduct a randomized controlled of the refined mHealth intervention.

DETAILED DESCRIPTION:
Aim 1. Develop an evidence and theory based WASH mHealth intervention for households in areas with confirmed cholera patients in Dhaka, Bangladesh through formative research

1. Conduct formative research through in-depth interviews, focus group discussions, and intervention planning workshops with caregivers and household members of young children, and government officials to identify perceptions of WASH behaviors and to inform the development of intervention materials.
2. Pilot the WASH mHealth intervention in a subset of households, and revise according to feedback.

Aim 2: Evaluate the effectiveness of the developed WASH mHealth intervention in increasing WASH behaviors and reducing fecal contamination on hands and in stored drinking water by conducting a RCT

1. Recruit and prospectively follow for 12 months 120 households (600 participants, 4 per household) with a child under five years of age assigned to one of two study arms (60 households per arm). The first arm will receive the CHoBI7 mHealth program (CHoBI7 mHealth program Arm) and the second arm will serve as a Control Arm and only receive a general message on oral rehydration solution (ORS).
2. Compare the 2 study arms using structured observation of handwashing with soap at stool and food related events, unannounced spot checks of the presence of soap in the cooking and latrine areas of the household, and fecal coliform counts on caregiver hands and in stored drinking water.

ELIGIBILITY:
Inclusion Criteria:

* At least one household member must report ownership of an active mobile phone in their possession on the day of enrollment

Exclusion Criteria:

* Household has a tap or basin with running water inside their home.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Marie George, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Households
Groups:
- CHoBI7 mHealth Program Arm: The first arm will receive the CHoBI7 mHealth program and a general message on oral rehydration solution (ORS) (CHoBI7 mHealth program Arm) .
  CHoBI7 mHealth program Arm: The investigators will start delivery of this intervention with a pictorial module delivered in the home during two 30 minute visits on cholera transmission and prevention after enrollment. Participants will be provided a handwashing station, a covered water vessel, and chlorine tablets. Participants will then receive the CHoBI7 WASH mHealth program voice and text messages on handwashing with soap and water treatment bi-weekly.
  general message on oral rehydration solution (ORS): general message on oral rehydration solution (ORS)
- Standard Recommendation Arm: The second arm participants will serve as a Control Arm and only receive a general message on oral rehydration solution (ORS).
  general message on oral rehydration solution (ORS): general message on oral rehydration solution (ORS)
Period: Overall Study
Arm/Group | CHoBI7 mHealth Program Arm | Standard Recommendation Arm
Started | 138; 39 Households | 146; 34 Households
Completed | 138; 39 Households | 146; 34 Households
Not Completed | 0; 0 Households | 0; 0 Households

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHoBI7 mHealth Program Arm | Standard Recommendation Arm | Total
Number analyzed (Participants) | 138 | 146 | 284
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 63 | 58 | 121
  Between 18 and 65 years | 75 | 88 | 163
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (15) | 24 (17.5) | 21 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 77 | 149
  Male | 66 | 69 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 138 | 146 | 284
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Bangladesh | 138 | 146 | 284

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Reported Handwashing With Soap at Stool and Food Related Events
Description: Handwashing with soap measured by 5-hour structured at the following food and stool related events in the household: (1) after using the toilet; (2) after cleaning a child's anus; (3) before eating; (4) before feeding a child; and (5) before preparing food.
Time Frame: 1 month, 3 months
Population: Participants that were available are reported
Measure: Count of Participants; unit: Participants
Arm/Group | CHoBI7 mHealth Program Arm | Standard Recommendation Arm
Number analyzed (Participants) | 138 | 146
Participants
  1 month: number analyzed (Participants) | 66 | 34
  1 month | 37 | 4
  3 months: number analyzed (Participants) | 62 | 46
  3 months | 27 | 10

2. Primary Outcome: Post Intervention Chlorine Concentration in Drinking Water
Description: Free available chlorine in stored household drinking water >0.2 mg/L
Time Frame: 7 Days after enrollment
Measure: Number; unit: Water samples with chlorine >0.2 mg/L
Units Other Than Participants: Household water samples
Arm/Group | CHoBI7 mHealth Program Arm | Standard Recommendation Arm
Number analyzed (Participants) | 138 | 146
Number analyzed (Household water samples) | 39 | 34
Water samples with chlorine >0.2 mg/L | 23 | 0

3. Secondary Outcome: Percentage of Diarrheal Events
Description: Participants will be asked if they have had diarrhea in the past week at the follow-up visits during the 3 month surveillance visit. Percentage of diarrheal events is reported.
Time Frame: Up to 3 months
Population: Individuals with clinical surveillance data available from follow-up visits during the 3 month-surveillance period
Measure: Mean (95% Confidence Interval); unit: percentage of diarrheal events
Groups:
- CHoBI7 mHealth Program Arm: The first arm will receive the CHoBI7 mHealth program and a general message on oral rehydration solution (ORS) (CHoBI7 mHealth program Arm) .
  CHoBI7 mHealth program Arm: We will start delivery of this intervention with a pictorial module delivered in the home during two 30 minute visits on cholera transmission and prevention after enrollment. Participants will be provided a handwashing station, a covered water vessel, and chlorine tablets. Participants will then receive the CHoBI7 WASH mHealth program voice and text messages on handwashing with soap and water treatment bi-weekly.
  general message on oral rehydration solution (ORS): general message on oral rehydration solution (ORS)
Arm/Group | CHoBI7 mHealth Program Arm | Standard Recommendation Arm
Number analyzed (Participants) | 80 | 76
percentage of diarrheal events | 11 [6 to 17] | 4 [1 to 7]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | CHoBI7 mHealth Program Arm | Standard Recommendation Arm
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/146
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/146
Other Adverse Events (participants affected / at risk) | 0/138 | 0/146

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT04816552/Prot_SAP_000.pdf